CLINICAL TRIAL: NCT03999346
Title: Opportunities and Limitations of Swiss Polytrauma Registry Data for Scientific Purposes- Registry Data for Scientific Purposes
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-01907; ch19Bless
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Trauma
Keywords: Swiss Polytrauma Registry; quality control; standardized identification procedures; data capture
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: retrospective analysis of the Swiss Trauma Registry data — retrospective analysis of protectively documented registry data based on data completeness, patient outcomes, patient characteristics

SUMMARY:
The aim of the analysis is an evaluation of the current performance of the Swiss Trauma Registry (STR) with respect to providing a reliable basis for (scientific) investigations on the management of trauma patients in Switzerland. The current project tries to address this question by considering central aspects of completeness and by exemplifying the use of the registry for research questions. The aim is to identify potential shortcomings of the registry.

ELIGIBILITY:
Inclusion Criteria:

* documentation in the STR
* Injury Severity Score (ISS) ≥ 16

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The data source for this project is the Swiss Trauma Registry with approx. 65 patients per year. Data will be extracted from the databank and transferred for analysis in anonymized form.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
analysis of data completeness | single time point assessment at baseline
  The STR comprises patient data starting from preclinical management, resuscitation, hospitalization and discharge data as well as data considering 28-day mortality, long-term outcome and cost. The founders agreed on a total of 98 items for analyses. All data sets will be evaluated for completeness of the 98 data points (items).
rate of 28 day survival | single time point assessment at baseline
  analysis of patient outcome: rate of patients' 28 day survival
length of hospital stay | single time point assessment at baseline
  analysis of patient outcome: length of hospital stay (days)
rate of patients receiving intensive care treatment | single time point assessment at baseline
  analysis of patient outcome: rate of patients receiving intensive care treatment
rate of patients returning to the previous living situation | single time point assessment at baseline
  analysis of patient outcome: rate of patients returning to the previous living situation

SECONDARY OUTCOMES:
cost of maintenance of the register | single time point assessment at baseline
  analysis of how many pro-rata salary per cent annually are specifically invested in the maintenance of the register

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Bless, Dr. med, Principal Investigator — Department Orthopedic and Trauma Surgery, University Hospital Basel
Locations (1):
- Department of Orthopaedics and Trauma Surgery (DOTS)., Basel, Switzerland